CLINICAL TRIAL: NCT00719823
Title: Maraviroc Compassionate Use
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4001068
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Maraviroc Compassionate Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 150mg, 300 mg or 600 mg twice daily administered orally with or without food in combination with other antiretroviral agents. The recommended dose of Maraviroc differs based on concomitant medications due to drug interactions as outlined in the Prescribing Information.

SUMMARY:
The objective of this study is to provide Maraviroc on a compassionate use basis to antiretroviral treatment experienced patients infected with CCR5-tropic HIV-1 with urgent unmet medical needs and who, in the opinion of the physician, require Maraviroc to form a viable regimen.

DETAILED DESCRIPTION:
This study was cancelled prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 16 years old with prior extensive treatment experience with limited further options in need of maraviroc to constitute an effective HIV-1 treatment regimen.
* Have only CCR5-tropic HIV-1 virus
* CD4+ cell count < 200 cells/mm3

Exclusion Criteria:

* CXCR4- or dual/mixed-tropic HIV-1 virus
* Patients who in the opinion of investigator are unlikely to derive benefit from maraviroc as a result of severity of illness
* Patients who are pregnant or breast feeding an infant or planning to become pregnant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Safety analysis will include all subjects who receive at least one dose of study drug | Two Years

SECONDARY OUTCOMES:
Safety analysis will include all subjects who receive at least one dose of study drug | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001068&StudyName=Maraviroc%20Compassionate%20Use